CLINICAL TRIAL: NCT06804187
Title: Identifying the Mechanisms of Gut-brain Axis to Sweet Sensing in Patients With Type 2 Diabetes Using Neuroimaging Techniques
Brief Title: Sweet Sensing in Type 2 Diabetes
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 24008
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Prediabetes
Keywords: sweet sensitivity; Type 2 diabetes; pre diabetes; sweet preference; sugar craving; taste receptors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Glucose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — blood samples will be taken and will check for glucose, HbA1c, c-peptide, insulin, 3-OMG and GLP-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Type 2 diabetes group: Inclusion criteria right or left handed age between 18-60 years HbA1c >48 mmol/mol duration of diabetes less than 10 years only for those who are treated with metformin
  excluding those with neurological disorder, gastrointestinal disorders, current pregnancy or breast feeding, on medications which can alter taste perception, current smokers, allergy to sugar, those who has contraindication to MRI, those who cannot lie flat, those who have taken part in research projects within the last 3 months
- Prediabetes group: Inclusion criteria right handed individuals age between 18-60 years HbA1c between 42-48 mmol/mol, diagnosis of pre-diabetes not less than 3 years only for those who are treated with metformin
  excluding those with neurological disorder, gastrointestinal disorders, current pregnancy or breast feeding, on medications which can alter taste perception, current smokers, allergy to sugar, those who has contraindication to MRI, those who cannot lie flat, those who have taken part in research projects within the last 3 months
- Healthy group: Inclusion criteria right or left handed individuals age between 18-60 years HbA1c </=42 mmol/mol only for those who are treated with metformin
  excluding those with neurological disorder, gastrointestinal disorders, current pregnancy or breast feeding, on medications which can alter taste perception, current smokers, allergy to sugar, those who has contraindication to MRI, those who cannot lie flat, those who have taken part in research projects within the last 3 months

SUMMARY:
Diabetes is a global challenge and the number of people affected by diabetes is expected to rise to 5.5 million by 2030, of which 90% are type 2 diabetes (T2D). Habitual high consumption of sugars is an important risk factor in the development, and progression, of type 2 diabetes (T2D). Several studies have now shown that individuals with T2D have reduced lingual sweet taste sensation and this in turns increases their sugar intake to achieve the same hedonic reward values compared to the healthy population. This subsequently will lead to development of diabetes or worsening of the blood sugar control.

Phase 1 of our study aims to identify the alterations in oral sweet taste sensitivity in individuals with type 2 diabetes and assess whether this is linked to sweet preference and habitual sugar consumption. In phase 2, we will use functional magnetic resonance imaging (MRI), a powerful technique used widely for diagnosing disease and investigating physiological and pathological process, to investigate whether diabetes or prediabetes status modulates activation of taste and reward-related brain responses to lingual sweet taste stimulation. Phase 3 will be investigating the reward-related brain responses to gut taste stimulation using functional MRI.

These new data will reveal the central mechanisms of sweet sensing in different status of diabetes and this will help develop novel treatment targets to improve metabolic and vascular outcomes in individuals with prediabetes or T2D.

ELIGIBILITY:
Inclusion Criteria:

* General Eligibility Criteria

  * For T2D: Confirmed Type 2 Diabetes Mellitus (HbA1c>48 mmol/mol (6.5%) and managed by the anti-diabetic drug metformin alone diagnosed within the last 10 years
  * For Prediabetes: HbA1c 42-48 mmol/mol and no less than 3 years since diagnosis
  * Non-diabetes who had HbA1c screened at their GP in the last 12 months: HbA1c≤42mmol/mol

Phase 1

Inclusion criteria:

Adults aged between 18 -60 years with type 2 diabetes or healthy individuals who had HbA1c checked within the last 12 months. Healthy volunteers who did not have HbA1c screened at their GP will be offered an opportunistic screening blood test.

Phase 2 and 3:

Inclusion criteria:

right-handed adults between 18- 60 years with type 2 diabetes, pre-diabetes and healthy individuals who had HbA1c checked within the last 12 months. Healthy volunteers who did not have HbA1c screened at their GP will be offered an opportunistic screening blood test.

Exclusion Criteria:

* Phase 1 exclusion criteria

  1. Current pregnancy or breastfeeding
  2. Current treatment with insulin or any other diabetic medications apart from metformin
  3. History of neurological, gastrointestinal injury or disease
  4. Any medication that is known to alter taste perception
  5. Smokers

Phase 2 and 3 exclusion criteria

1. individuals with Neurological or gastrointestinal disorders (IBD/ IBS)
2. those who have contraindications to MRI including metal implants
3. those who are unable to lie flat
4. smokers
5. those who have taken part in research projects within the last 3 months (projects involving administering a drug, invasive procedure i.e. venepuncture >50 ml, endoscopy, or exposure to ionising radiation)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will be inviting potential participants from primary care team and also healthy volunteer from the university campus or to the public by displaying poster around the campus and health facilities.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To assess the sensitivity and preference of lingual sweet taste in individuals with T2D, and those without T2D to evaluate how this is impacted by habitual sugar consumption. | December 2024 to December 2026
To compare brain responses to lingual sweet sensing in individuals with prediabetes and T2D, and those without prediabetes or T2D, and their association with habitual sugar consumption. | from Dec 2024 to Dec 2026

SECONDARY OUTCOMES:
To determine how brain responses to intestinal sweet sening predict the rate of intestinal glucose absorption. | Feb 2025 to Dec 2026

CONTACTS AND LOCATIONS:
Overall Officials: Sally Eldeghaidy, BSc, MSc, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, East Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are not planning to share individual participant data but will publish in scientific papers and conferences with the overall results.